# **Informed Consent Form**

## **Study Title:**

Effects of Two Different Natural Nutritional Supplements on Anaerobic Performance and Muscle Oxygenation in U-19 Football Players

## **Principal Investigator:**

Dr. Melike Nur EROGLU Department of Sports Sciences, Sakarya University of Applied Sciences

#### **Contact Information:**

Phone: +905384982024

Email: melikeeroglu@subu.edu.tr

Date:

July 01 2024

## Informed Consent Form

#### 1. Purpose of the Study

This study aims to investigate the effects of two different natural nutritional supplements on anaerobic performance and muscle oxygenation in young male football players. Various performance and physiological parameters will be measured during the study.

#### 2. Study Procedures and Duration

You will be asked to attend three laboratory visits. During two of these visits, you will consume one of the two natural supplements or a placebo in a randomized, double-blind, crossover design. There will be a 7-day washout period between these sessions. The total study duration is approximately 3 weeks.

#### 3. Participant Eligibility

You are eligible to participate if you:

- Are a healthy male aged 18 years or older
- Engage in resistance exercise at least 3 times per week
- Have at least 5 years of football training experience

You are not eligible if you:

- Have contraindications to Wingate exercise testing
- Have cardiometabolic disease
- Are currently using ergogenic supplements
- Smoke tobacco

#### 4. Study Procedures

At each testing session, you will:

- Perform a Wingate anaerobic test on a cycle ergometer
- Consume one of the two natural nutritional supplements or placebo 2.5 hours before exercise
- Undergo measurements including muscle oxygenation, blood lactate, blood glucose, blood pressure, heart rate, and perceived exertion

You will be asked to maintain your regular diet and exercise habits, with some restrictions 24-48 hours before testing (such as avoiding nitrate-rich foods, caffeine, alcohol, and intense exercise).

#### 5. Blinding and Disclosure

To maintain the integrity of the study, neither you nor the investigators will know which supplement you are receiving during each session. This information will be disclosed to you only after the study is fully completed.

#### 6. Risks and Discomforts

The study involves physical exertion which may cause temporary fatigue or muscle soreness. The supplements used are natural and generally safe, but mild side effects such as gastrointestinal discomfort may occur.

#### 7. Benefits

Although there may be no direct benefit to you, the findings may help improve nutritional strategies to enhance athletic performance.

#### 8. Confidentiality

Your personal information will be kept confidential and only used for research purposes. Results will be reported anonymously.

#### 9. Voluntary Participation and Withdrawal

Participation is voluntary. You may withdraw at any time without any negative consequences.

#### 10. Questions and Contacts

If you have any questions, please contact the principal investigator at [+905384982024] or [melikeeroglu@subu.edu.tr].

#### **Consent Statement:**

I have read and understood the above information. I have had the chance to ask questions. I voluntarily agree to participate in this study under the conditions described.

| Participant Name (Pi | rinted): |
|----------------------|----------|
|----------------------|----------|

| Participant Signature: |
|------------------------------|
| Date: |
| Investigator Name (Printed): |
| Investigator Signature: |
| Date: |